CLINICAL TRIAL: NCT06749262
Title: Inducing Variable Breathing Ratios During Walking to Improve Exercise Capacity in Patients With Chronic Obstructive Pulmonary Disease.
Brief Title: Inclined Versus Standard Exercise for COPD Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: F5337-R; I01RX005337-01A1 (Other Grant/Funding Number: VA)
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: pulmonary rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Interventional longitudinal study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Walking at Incline (Experimental): Subjects will walk on treadmill at slope equal to 60% of their peak heart rate as determined on baseline cardiopulmonary exercise test.
  Interventions: Other: walking on incline or walking at increasing speed for 36 visits
- Walking at Speed (Experimental): Subjects will walk on treadmill at speed equal to 60% of their peak heart rate as determined on baseline cardiopulmonary exercise test.
  Interventions: Other: walking on incline or walking at increasing speed for 36 visits

INTERVENTIONS:
Other: walking on incline or walking at increasing speed for 36 visits — Subjects will be prepared for data collection by wearing an exercise suit and obtaining height and body weight. Breathing sensors and foot switches will be worn to measure breathing and walking performance.

SUMMARY:
This study is designed to provide information regarding how to improve pulmonary rehabilitation for persons with chronic obstructive pulmonary disease (COPD). Pulmonary rehabilitation is an exercise program for COPD patients that is recommended and benefits some, but not all, patients. The question being studied in this trial is whether during an exercise program, walking on an incline might be better than walking on faster on a flat surface in training muscles so that patients might be less short of breath with exercise.

DETAILED DESCRIPTION:
Objective: The objective of this project is to determine the effect of a pulmonary rehabilitation program that utilizes inclined versus standard exercise to improve breathing and walking for individuals with COPD.

Research Design: Fifty-six patients with COPD (28 in each treatment group: inclined or standard rehabilitation) will be recruited through the VA Nebraska-Western Iowa Health Center clinics. Patients will be randomly assigned to either inclined or standard rehabilitation groups and participate in a 12-week pulmonary rehab program (3 sessions/ week). Potential research subjects will undergo a medical history exam & pulmonary function test at the Omaha VA, and a maximal cardiopulmonary exercise test (CPET) at the Nebraska Cardiac Pulmonary Rehab Center (Rehab Center). Only those that are cleared for participation by a physician will be enrolled.

Methodology: The study will be conducted at the Omaha VA and the Rehab Center. All subjects will be diagnosed with chronic obstructive pulmonary disease (COPD) with no other significant co-morbidities and screened for eligibility. Up to 108 patients may be consented and screened to achieve target enrollment of 58 subjects.

Enrolled participants will first complete a series of questionnaires that will be used as covariates in the analysis at the Rehab Center then proceed with their first rehab session.

The Q-stress system, connected to the participants while they walk on a treadmill, will be used to monitor participants' cardiovascular responses. The treadmill's speed and incline will be incrementally increased until the participants reach 60% of their maximal heart rate as determined by the CPET. For both the standard treadmill walking and incline walking, the goal is to achieve 30 minutes of walking at the 60% intensity without a break at the end of the 12 weeks. For the standard walking, subjects will walk at their preferred speed, on a 0% level surface of the treadmill. The treadmill speed will be incrementally enhanced by 0.05 meters per second each minute until the participant's heart rate attains 60% of the maximal heart rate recorded during the CPET. With the inclined treadmill walking group, participants will begin walking at a pace 20% below their preferred walking speed on a 2% incline, which will then be elevated by 0.5% each minute. Each session will last up to 50 minutes plus 5 minutes of warm-up and cool-down. After completing a session, interviews and questionnaires will be used to assess comfort, fatigue, and exercise intensity.

Outcome measures from the Q-stress system are respiratory flow pattern, dyspnea, dynamic hyperinflation, LRC ratio, total walking time and metabolic equivalence of task (METs).

Clinical relationship: COPD is a major health concern for the Department of Veterans Affairs. Current pulmonary rehabilitation programs do not consistently improve outcomes. Enhancing the effectiveness of these programs could significantly improve patient outcomes. The investigators hypothesize that inclined walking will reduce respiratory rate, dynamic hyperinflation, and dyspnea, thereby improving exercise capacity and quality of life for these patients. These findings can be incorporated into rehabilitation practices, reducing the disability linked to the disease and enhancing the overall health outcomes for Veterans.

ELIGIBILITY:
Inclusion Criteria:

* Veterans from all sex/gender, race, and ethnicity will be recruited
* All subjects will undergo post-bronchodilator spirometry and be clinically stable
* All subjects must have documented FEV1/FVC ratio of <0.7, and between 30% to 80% FEV1% predicted
* If subjects have non-qualifying spirometry, they will not be screened further
* Subjects with qualifying spirometry will be screened further
* Potential subjects must have a BMI of less than 35 kg/m2 and must be free from co-morbidities that may affect walking patterns

  * e.g., peripheral arterial disease, diabetes, low back pain

Exclusion Criteria:

* Confounding effects such as neurological, musculoskeletal, or metabolic disease
* Subjects taking medications that alter mood or metabolic demand will be excluded
* All potential subjects must be cleared for participation by a physician after undergoing a cardiopulmonary exercise test
* Require an O2 mask during rest or activity

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-09-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Respiratory rate | During each session of Exercise up to 12 weeks
  Respiratory rate will be analyzed using motion capture markers on the chest. With custom computer code, the markers will be identified to model a sphere. The volume of the sphere will be recorded over time. As the volume increases and decreases, respiratory flow will be identified, and respiratory rate can be calculated.
Dyspnea | During each session of Exercise up to 12 weeks
  Perceived dyspnea: Breathlessness will be measured based on a 0 to 10-point Borg scale at the end of the treadmill trials. 0 on scale is no breathlessness and 10 is maximal breathlessness
Dynamic hyperinflation | During each session of Exercise up to 12 weeks
  Dynamic hyperinflation will be assessed by inspiratory capacity through pre- and post-walking trial resting spirometry. Dynamic hyperinflation will be considered to be present when inspiratory capacity values decrease after walking trials when compared to resting values.
Total walking time | During each session of Exercise up to 12 weeks
  Total walking time will be assessed by measuring the time that each participant walks during an exercise session

OTHER OUTCOMES:
Locomotor respiratory coupling (LRC) | During each session of Exercise up to 12 weeks
  The investigators will measure synchronized respiratory cycles using RIP bands and walking cycles using SMTEC footswitch system (Sport & Medical Technologies SA, Nyon, Switzerland) to detect gait events. LRC is often quantified as frequency coupling. Frequency coupling refers to how many heel strikes occur within a single cycle of respiration (one inhalation to the next); it is usually counted in integer or half-integer ratios, measured using discrete relative phase between walking (heel strikes) and breathing rhythms time series. Discrete relative phase values between 0º-360º have a 1:1 relationship, 360º-720º have a 2:1 relationship, 720º-1080º have a 3:1 relationship, and so on. Half-integer couplings (expressed as 3:2, 5:2, 7:2, etc.) exist when the frequency alternates between two integers. The range of ratios and the percentage of time each ratio is utilized will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Kristina L Bailey, Principal Investigator — Omaha VA Nebraska-Western Iowa Health Care System, Omaha, NE
Locations (1):
- Omaha VA Nebraska-Western Iowa Health Care System, Omaha, NE, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No